CLINICAL TRIAL: NCT06291675
Title: Long-term Observational Study to Investigate the Effect of Gender-affirming Hormone Therapy (GAHT) on Heart Function Parameters, Heart, Liver and Pancreatic Fat Content as Well as the Insulin System and the Psychological Impact of GAHT
Brief Title: Gender-Affirming Hormone Therapy and Its Impact on Myocardial Mass and Cardiac Function, Heart, Liver and Pancreatic Fat Content
Status: Recruiting | Type: Observational
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Alexandra Kautzky-Willer, Principal Investigator, Medical University of Vienna
Other Study IDs: 2083/2022
Record Dates: First submitted 2024-01-25; First posted 2024-03-04 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: Gender Dysphoria; Hormone Therapy Induced Morphologic Change
MeSH Terms: conditions — Gender Dysphoria

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Transgender women: Transgender women included in this study receive estrogen, either transdermally (Estrogel-Gel®, Estradot® or Estramon®) or orally (Estrofem®). If needed, the treatment can be supplemented by cyproterone acetate (Androcur®), and/or an alpha-5-reductase inhibitor (Finasterid Actavis/Arcana/Aurobindo®). The GAHT of our probands is prescribed and managed independently of the study, and the study has no effect on the treatment.
  Interventions: Drug: gender-affirming hormone therapy
- Transgender men: The cohort of transgender men are persons who receive testosterone either intramuscularly (Nebido®) or transdermally (Testogel® or Testavan®). The GAHT of our probands is prescribed and managed independently of the study, and the study has no effect on the treatment.
  Interventions: Drug: gender-affirming hormone therapy

INTERVENTIONS:
Drug: gender-affirming hormone therapy — We are not technically involved in the prescription of gender-affirming hormone therapy. We merely aim at observing effects of GAHT on MRI measured organ lipid content, myocardial mass and function.

SUMMARY:
Background: Gender affirming hormone therapy (GAHT) leads to profound changes in sex hormone levels, carrying a wide range of implications for major physiological processes in the body. GAHT has been shown to be associated with changes in cardiovascular parameters, the insulin system, body composition, and the psychological state. However, despite the fact that GAHT is usually a long-term intervention, the majority of the research concerns itself with an overall short duration of the therapy and the data on the mid- to long-term effects of GAHT is scarce.

Objectives: The study aims to investigate the effects of gender affirming hormone therapy on the cardiovascular risk profile, insulin system, body composition, various metabolic parameters, and the psychological state after 2, 5, and 10 years of the treatment.

Study design: The study is designed as an observational longitudinal monocentric study, which includes transgender men and transgender women who have been taking gender affirming hormone therapy during the past 2 years and took part in our pilot study. Our probands will undergo a magnetic resonance scan, extensive bloodwork, an oral glucose tolerance test, and a psychological self-assessment after 2, 5, and 10 years of the treatment.

Materials and methods: The magnetic resonance imaging and spectroscopy will be performed with a 3-Tesla magnetic resonance device. We will also perform an extensive blood analysis and an 75g- 2h oral glucose tolerance test. Additionally, the psychological state of the probands will be assessed with 3 questionnaires.

Study population: 30 transgender men 30 transgender women who participated in our pilot study and have been taking the gender affirming hormone therapy for the past 2 years.

Relevance and implications of the study: The majority of previous research has focused on the short-term effects of gender affirming hormone therapy. Contrastingly, our study aims to focus on the effects of hormone therapy at 2, 5 and 10 years after the beginning of the treatment. Moreover, our study group utilizes measurements of myocardial, hepatic, and pancreatic fat content as well as an MR-assisted measurement of cardiac function, which is a topic that has not been present in research into the effects of gender affirming hormone therapy outside of our pilot study.

DETAILED DESCRIPTION:
Background Gender affirming hormone therapy is a treatment used by many transgender individuals aiming for physical transition. During this treatment, the endogenous production of sex hormones is reduced, and they are supplemented by the sex hormones of the gender with which the person identifies. These profound changes in the hormonal profiles of transgender people have been shown to be associated with changes in cardiovascular parameters, the insulin system, body composition, and the psychological state.

In the case of transgender men under GAHT, the treatment seems to be associated with the development of a less favorable, more atherogenic lipid profile, with an increase in triglycerides and low-density lipoprotein (LDL) levels, while also experiencing a decrease in high-density lipoprotein (HDL). On the other hand, transgender women under GAHT seem to develop higher levels of triglycerides, with little to no changes in LDL and HLD levels. Additionally, GAHT seems to have an effect on body composition - in transgender men, GAHT is associated with a decrease in fat mass, on the other hand, in transgender women GAHT is connected to an increase in total body fat. These changes do not seem to be associated with a significant change in the visceral fat mass in either group (Klaver et al., 2022).

Despite the documented effects of GAHT on cardiovascular risk factors, it is still not entirely clear whether these effects are significant enough to cause significant changes in cardiovascular morbidity and mortality. However, the prior findings suggest that transgender women have a higher risk of suffering an ischemic stroke or a myocardial infarction compared to cisgender women, while there is no consistent evidence documenting an increase of cerebrovascular and cardiovascular disease transgender men compared to cisgender men.

The research into changes in glucose homeostasis has not delivered conclusive long-term findings so far. Nevertheless, there is a documented tendency towards a slight worsening of insulin sensitivity in transgender women, while the effects of GAHT on insulin resistance in transgender men are associated with either no change or a small improvement.

Gender affirming hormone treatment also seems to have an impact on the psychological and cognitive state of the patients, for example, it has been brought into connection with an alleviation of depressive symptoms. Furthermore, there are documented morphological and functional changes in the brains of people taking GAHT. These changes might be accompanied by changes in neuropsychological processes, including, for example, emotional regulation. Additionally, there is a lack of data on the possible changes in executive function in transgender people, especially in regard to longitudinal changes under GAHT.

Long-term studies are still lacking in the realm of sequelae of GAHT. Thus, we aim at observing and investigating psychological and cardiovascular effects of GAHT in the long-term.

3.3. Study design The study is designed as a prospective longitudinal mono-centric observational study comparing cardiovascular and psychological effects of GAHT after 2, 5, and 10 years of GAHT with the patient's status before GAHT. We aim at enrolling all participants of our pilot study (EK 1629/2017) who started GAHT in the last two years and have, thus, completed the psychological assessments before the start of GAHT.

At each visit, our probands will undergo a magnetic resonance scan, an oral glucose tolerance test, as well as an extensive blood analysis and an assessment of the anthropometric parameters. Additionally, the patient history and self-assessment with standardized psychological tests will be performed at each visit. The study will include 3 separate study visits, after 2, 5, and 10 years of treatment.

3.4. Subject section Our study aims to enroll transgender probands who took part in our pilot study. 30 transgender women and 30 transgender men will be recruited from the pool of participants in the previous pilot study (EK 1629/2017). The study will include transgender participants between 18 and 99 years of age, who have been taking gender affirming hormone therapy for the past 2 years. The study will not include a placebo group or a control group, and it will not interfere with the gender affirming hormone therapy in any way regarding composition and time course of the treatment.

3.5. Hormones/treatment protocols The gender affirming hormone treatment protocols of our probands are based on the protocols as used by the outpatient clinic specializing in gender affirming hormone treatment at the Departments of Endocrinology and Metabolism and Gynecology and Obstetrics of the Vienna General Hospital/Medical University of Vienna. The GAHT of our probands is prescribed and managed independently of the study, and the study has no effect on the treatment.

Transgender women included in this study receive estrogen, either transdermally (Estrogel-Gel®, Estradot® or Estramon®) or orally (Estrofem®). If needed, the treatment can be supplemented by cyproterone acetate (Androcur®), and/or an alpha-5-reductase inhibitor (Finasterid Actavis/Arcana/Aurobindo®).

Transgender men included in this study receive testosterone either intramuscularly (Nebido®) or transdermally (Testogel® or Testavan®). If necessary, the treatment might be supplemented by lynestrenol (Orgametril®).

Furthermore, the treatment in both cohorts can, if necessary, be complemented by GnRH analogues, such as triptorelin acetate (Decapeptyl® or leuprorelin acetate every 3 months (Trenantone®).

4. Methods and materials All measurements and assessments will be performed after an overnight fast of minimum 8 hours.

4.1. Magnetic resonance imaging and spectroscopy Magnetic resonance spectroscopy is a possible non-invasive method for quantifying ectopic accumulation of lipids. Intramyocardial, hepatic and pancreatic fat content, as well as subcutaneous and visceral fat and parameters of cardiac function will be measured using magnetic resonance imaging and magnetic resonance spectroscopy in a 3-Tesla Magnetom PrismaFit magnet (Siemens Healthliners, Erlangen, Germany). Magnetic resonance imaging and spectroscopy will be conducted in accordance with established protocols, which have previously been used in our pilot study.

For the measurements of visceral and subcutaneous adipose tissue, T1-weighted visualizations in an axial slice in the L2/L3 area will be used. Pancreatic fat content will be quantified following a protocol similar to one previously published by Al-Mrabeh et al., which utilizes fat fraction images derived from multi-echo Dixon imaging sequences. Additionally, hepatic and myocardial fat content will be assessed by short time single voxel spectroscopy and electrocardiogram-gated spectroscopy respectively.

4.2. Bloodwork and oral glucose tolerance test Our study will include extensive bloodwork with an analysis of metabolic parameters, cardiovascular risk factors, and various other biomarkers. After the initial blood draw, an oral glucose tolerance test will be performed. After taking the baseline sample, the probands will be asked to ingest 75 grams of glucose dissolved in 200ml of water. Subsequently, blood samples will be taken 30, 60, 90, and 120 minutes after the glucose ingestion, and the concentrations of glucose, insulin and c-peptide will be measured from the samples. For the repeated blood draws, an intravenous cannula will be placed preferably into the cubital vein. The measured concentrations will be used to calculate the surrogate markers for insulin sensitivity/insulin resistance (HOMA-IR, Matsuda-Index, Stumvoll first and second phase indices).

The samples will be analyzed at an ISO 9001 certified laboratory of the Vienna General Hospital, according to the established protocols of the Institute of Laboratory Medicine. Adiponectin and betatrophin will be measured by human ELISA kits from the company Biovendor.

4.3. Assessment of psychological and cognitive state The patients will be asked to fill out 3 standardized questionnaires for an assessment of their psychological and cognitive state. Depressive symptoms will be evaluated by the Becks depression inventory self-rating scale (BDI-II) which consists of 21 items. Emotion control, processing, avoidance, and repression will be quantified with the 25-item Emotional Process Scale (EPS-D). Additionally, the Trier personality questionnaire (TPF) will be used for evaluating psychological wellbeing. The questionnaires will be handed to the probands during the OGTT and are intended to be filled out during the waiting times between the blood draws. The questionnaires will then be analyzed by the psychologist involved in this study, Mag. Maria-Christine Mautner. Should a patient show an increased risk for endangerment of self or others in a psychological questionnaire, the patient will be informed and they will immediately be referred to the crisis intervention center of the Vienna General Hospital.

4.4. Other parameters Blood pressure and heart rate will be measured with an OMRON 705 device on the left arm after a minimum of 10 minutes at rest. Weight will be measured on calibrated electronic scales (SECA 877/888) to the nearest 0,1 kg wearing light clothes and no shoes. The body mass index will be calculated from the measured weight and self-reported height. Waist circumference will be measured at the midpoint between the lower border of the rib cage twice, and the average of the two measurements will be recorded.

5. Statistical and data analysis After the completion of the study, we will have data at several time points. To be exact, we will have measured systolic and diastolic heart function, hepatic, pancreatic, and myocardial fat content, subcutaneous to visceral fat ratio, variables on the functionality of the insulin system, information on depression, emotion and behavioral control as well as adiponectin and betatrophin concentration after 2, 5, and 10 years of the treatment. Initially, the data will be tested for normal distribution using the Kolmogorov-Smirnov and Shapiro-Wilks tests. If necessary, logarithmic transformation will be performed. The comparisons between the different time points will be performed using a repeated measure ANOVA. Possible correlations will be tested using Pearson's or Spearman's correlation coefficients. The data will also be presented as mean ± standard deviation, or median ± interquartile range, as appropriate. The level of significance will be set at α < 0,05. The data will be tested using the IBM SPSS Statistics Software (Version 29, IBM, New York, USA).

6. Ethical section The study will be performed under the Declaration of Helsinki (1964) and the Good Clinical Practice guidelines.

The gender affirming hormone therapy of the probands is clinically indicated and completely independent from our study. The study does not influence the composition, start, duration, or end of the treatment. All subjects will receive a thorough patient information and will sign informed consent forms prior to the inclusion in the study. The probands will be able to withdraw from the study at any time. Additionally, the study team has the right to remove participants from the study if the exclusion criteria have been met, or if the participation in the study is not in the best interest of the proband.

No significant side effects are expected from any of the procedures included in the study. In the case of possible concerning findings made during the examinations, the probands will be offered a consultation and will be referred to the appropriate diagnostic or therapeutic procedures. Should a patient show an increased risk for endangerment of self or others in a psychological questionnaire, they will immediately be referred to the crisis intervention center of the Vienna General Hospital.

7. Human resources, study sites, cooperations The proposed study will be conducted at the Department of Endocrinology and Metabolism (head: Univ. Prof. Dr. Alexandra Kautzky-Willer; collaborators: Dr. Carola Deischinger, Dr. Jürgen Harreiter, Dr. Dorota Sluková, Mag. Maria-Christine Mautner, Dr. Lana Kosi-Trebotic), the Department of Obstetrics and Gynecology, Division of Gynecologic Endocrinology and Reproductive Medicine, Unit for Gender Identity Disorder (Ulrike Kaufmann, MD) of the Medical University of Vienna / General Hospital of Vienna. and the High Field MR Centre (collaborators: Ivica Just, MSc PhD; Mag. Radka Klepochova, PhD; Assoc. Prof. Dr. Martin Krššák).

8. Relevance and implications of the study Despite the fact that gender affirming hormone therapy is usually a long-term intervention, the majority of the research into its effects concerns itself with only the short-term effects. Thus, there is an obvious need for more longitudinal research into the longer-term effects of GAHT in order to assess the potential effects of gender affirming hormone therapy more appropriately and to provide better personalized patient care. Our study aims to provide more insight into the mid- to long-term effects of gender affirming hormone treatment in both transgender women and transgender men.

Furthermore, apart from our pilot study, we are not aware of a study including MRI and MRS-assisted measurements of SAT, VAT, hepatic, pancreatic and myocardial fat content and cardiac function in people taking gender affirming hormone therapy.

ELIGIBILITY:
Inclusion Criteria:

* participation in our pilot study

  * ongoing gender affirming hormone therapy during the last 2 years
  * willingness and competence to sign the informed consent form.

Exclusion Criteria:

* age < 18 years

  * non-MRI conditional implants, grafts, and/or devices
  * non-MRI conditional tattoos
  * claustrophobia
  * current substance abuse
  * pregnancy
  * failure to comply with the study protocol and/or not following the instructions of the study team.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Transgender men and transgender women are selected according to their experienced gender
Study Population: Our study aims to enroll transgender probands who took part in our pilot study. 30 transgender women and 30 transgender men will be recruited from the pool of participants in the previous pilot study (EK 1629/2017). The study will include transgender participants between 18 and 99 years of age, who have been taking gender affirming hormone therapy for the past 2 years. The study will not include a placebo group or a control group, and it will not interfere with the gender affirming hormone therapy in any way regarding composition and time course of the treatment.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2023-03-03 (Actual); Primary Completion 2027-03-03 (Estimated); Study Completion 2033-03-03 (Estimated)

PRIMARY OUTCOMES:
Myocardial mass | after 2, 5 and 10 years of gender-affirming hormone therapy
  to examine the effects of gender affirming hormone treatment on myocardial mass (in g/m³)
Cardiac function - LVEF | after 2, 5 and 10 years of gender-affirming hormone therapy
  to examine the effects of gender affirming hormone treatment on left-ventricular ejection fraction (in %) (LVEF) using MR-assisted measurements
cardiac function - cardiac output index | after 2, 5 and 10 years of gender-affirming hormone therapy
  to examine the effects of gender affirming hormone treatment on cardiac output index (in L/min/m²) using MR-assisted measurements
Organ lipid content | after 2, 5 and 10 years of gender-affirming hormone therapy
  to examine the effects of gender affirming hormone treatment on hepatic, pancreatic, and myocardial fat content after 2, 5, and 10 years of the treatment using MR-assisted measurements
Subcutaneous to visceral fat ratio | after 2, 5 and 10 years of gender-affirming hormone therapy
  to examine the effects of gender affirming hormone treatment on subcutaneous to visceral fat ratio after 2, 5, and 10 years of the treatment using MR-assisted measurements

CONTACTS AND LOCATIONS:
Overall Officials: Alexandra Kautzky-Willer, Prof, MD, Principal Investigator — Medical University of Vienna
Locations (1):
- Chiari Stoffwechselambulanz, Medical University of Vienna, Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: Undecided
Maybe anonymized patient data might be shared with other European researchers from the ENIGI network (if adequate ethics statement is available)